CLINICAL TRIAL: NCT01155778
Title: A Phase I/II Safety, Tolerability, Ascending Dose and Dose Frequency Study of Recombinant Human Heparan N-Sulfatase (rhHNS) Intrathecal Administration Via an Intrathecal Drug Delivery Device in Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Brief Title: Safety, Tolerability, Ascending Dose and Dose Frequency Study of rhHNS Via an IDDD in MPS IIIA Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-SAN-055; 2009-015984-15 (EudraCT Number)
Record Dates: First submitted 2010-06-24; First posted 2010-07-02 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Mucopolysaccharidosis (MPS)
Keywords: Mucopolysaccharidosis (MPS) IIIA; Recombinant Human Heparan N-Sulfatase (rhHNS); Sanfilippo Syndrome Type A (MPS IIIA); Lysosomal Storage Disease (LSD); Intrathecal Drug Delivery Device (IDDD)
MeSH Terms: conditions — Mucopolysaccharidoses; Mucopolysaccharidosis III; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 mg rhHNS (Experimental): 10 mg monthly via an IDDD (every 28 [±7 days]) for a total of 6 months
  Interventions: Biological: Recombinant human heparan N-sulfatase (rhHNS)
- 45 mg rhHNS (Experimental): 45 mg monthly via an IDDD (every 28 [±7 days]) for a total of 6 months
  Interventions: Biological: Recombinant human heparan N-sulfatase (rhHNS)
- 90 mg rhHNS (Experimental): Given IDDD as a 45 mg dose every 14 [±2 days] for a monthly total of 90 mg for 6 months
  Interventions: Biological: Recombinant human heparan N-sulfatase (rhHNS)

INTERVENTIONS:
Biological: Recombinant human heparan N-sulfatase (rhHNS)

SUMMARY:
Sanfilippo syndrome, or Mucopolysaccharidosis (MPS) III, is a rare lysosomal storage disease (LSD) caused by loss in activity of 1 of 4 enzymes necessary for degradation of the glycosaminoglycan (GAG) heparan sulfate (HS) in lysosomes. MPS IIIA results from deficiency of the enzyme heparan N-sulfatase (sulfamidase). MPS IIIA symptoms arise on average at 7 months of age, with the average age of diagnosis at 4.5 years for the majority of patients. The central nervous system (CNS) is the most severely affected organ system in patients with MPS IIIA, evidenced by deficits in language development, motor skills, and intellectual development. In addition, there are abnormal behaviors including but not limited to aggression and excess motor activity/hyperactivity that contribute to disturbances in sleep.Overall, individuals with MPS IIIA have a marked developmental delay and significantly reduced lifespan of 15 years of age on average.

The purpose of this study is to determine the safety and tolerability of rhHNS via ascending doses administered via an a surgically implanted intrathecal drug delivery device (IDDD) intrathecal (IT) route once monthly (or every two weeks) for 6 months in patients with MPS IIIA.

DETAILED DESCRIPTION:
No effective, disease-modifying therapies are currently approved as treatments for this devastating and disabling disease.

Shire Human Genetic Therapies (Shire HGT) is developing a sulfamidase enzyme replacement therapy (ERT)rhHNS for patients with MPS IIIA. recombinant human heparan-N-sulfatase (rhHNS) is being administered into the cerebrospinal fluid (CSF) via an surgically implanted intrathecal drug delivery device (IDDD), because when administered intravenously (IV) it does not cross the blood brain barrier (BBB).

This study is a multicenter, multiple-dose, dose escalation study designed to evaluate the safety, tolerability, and clinical activity of up to 3 dose levels (10mg,45mg and 90mg monthly for 6 months) of rhHNS administered via an IDDD in patients with Sanfilippo syndrome Type A ages greater than or equal to 3 years of age.

Patients who have completed all study requirements in this study will be invited to participate in an open-label extension study that will be designed to evaluate long term safety and clinical outcomes of intrathecal administration of rhHNS.

ELIGIBILITY:
Inclusion Criteria

Each patient had to meet the following criteria to be eligible for the study:

1. a.) Patients had a documented deficiency in sulfamidase enzyme activity of ≤10% of the lower limit of the normal range as measured in fibroblasts or leukocytes.

   AND either b or c b.) Patients had a normal enzyme activity level of at least 1 other sulfatase (to rule out multiple sulfatase deficiency) as measured in fibroblasts or leukocytes.

   c.) Patients had 2 documented mutations.
2. The patient was ≥3 years of age and had a developmental age ≥1 year.
3. Patients must have been medically stable, in the opinion of the Investigator, to accommodate the protocol requirements, including travel, assessments, and IDDD surgery, without placing an undue burden on the patient/patient's family.
4. The patient's parent(s) or legal guardian must have voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient, the patient's parent(s), or legal guardian. The patients, patient's parents or legal guardian's consent and patient's assent as appropriate, must have been obtained.

Exclusion Criteria

Patients who met any of the following criteria were excluded from the study:

1. The patient had significant non-MPS IIIA related CNS impairment or behavioral disturbances that would confound the scientific integrity or interpretation of study assessments, as determined by the investigator.
2. The patient had MPS IIIA behavioral-related issues, as determined by the investigator, that would have precluded performance of study neurocognitive and developmental testing procedures
3. The patient was pregnant, breast feeding, or was a female patient of childbearing potential who would not or could not comply with the use of an acceptable method of birth control such as condoms, barrier method, oral contraception, etc.
4. The patient was blind and/or deaf.
5. The patient had any known or suspected hypersensitivity to anesthesia or was thought to have an unacceptably high risk for anesthesia due to airway compromise or other conditions.
6. The patient or the patient's family had a history of neuroleptic malignant syndrome, malignant hyperthermia, or other anesthesia-related concerns.
7. The investigator may have chosen to exclude patients who have had complications resulting from prior lumbar punctures.
8. The patient had a CNS shunt.
9. The patient had skeletomuscular/spinal abnormalities or other contraindications for the surgical implantation of the IDDD.
10. The patient had a history of poorly controlled seizure disorder.
11. The patient was currently receiving psychotropic or other medications, which in the investigator's opinion, would have been likely to substantially confound test results and the dose and regimen of which cannot be kept constant throughout the study.
12. The patient could not sustain absence from aspirin, non-steroidal medications, or medications that affected blood clotting within 1 week prior to a relevant study related procedure (eg, device implantation if applicable), or had ingested such medications within 1 week before any procedures in which any change in clotting activity would have been deleterious.
13. The patient had received treatment with any investigational drug or a device intended as a treatment for MPS IIIA within the 30 days prior to, or during the study, or was enrolled in another study that involved an investigational drug or device (screening through safety follow-up contact).
14. The patient received a hematopoietic stem cell or bone marrow transplant.
15. The patient's parent(s), or patient's legal guardian(s) was/were unable to provide consent or the patient could not provide assent, as appropriate, due to, but not limited to, the inability to understand the nature, scope, and possible consequences of the study, or did not agree to comply with the protocol defined schedule of assessments.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2012-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Emma Children's Hospital, Academic Medical Center, Amsterdam, Netherlands
- St. Mary's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Jones SA, Breen C, Heap F, Rust S, de Ruijter J, Tump E, Marchal JP, Pan L, Qiu Y, Chung JK, Nair N, Haslett PAJ, Barbier AJ, Wijburg FA. A phase 1/2 study of intrathecal heparan-N-sulfatase in patients with mucopolysaccharidosis IIIA. Mol Genet Metab. 2016 Jul;118(3):198-205. doi: 10.1016/j.ymgme.2016.05.006. Epub 2016 May 10. PMID 27211612
- [Derived] King B, Marshall N, Beard H, Hassiotis S, Trim PJ, Snel MF, Rozaklis T, Jolly RD, Hopwood JJ, Hemsley KM. Evaluation of enzyme dose and dose-frequency in ameliorating substrate accumulation in MPS IIIA Huntaway dog brain. J Inherit Metab Dis. 2015 Mar;38(2):341-50. doi: 10.1007/s10545-014-9790-8. Epub 2014 Nov 25. PMID 25421091
- [Derived] Langford-Smith A, Wilkinson FL, Langford-Smith KJ, Holley RJ, Sergijenko A, Howe SJ, Bennett WR, Jones SA, Wraith J, Merry CL, Wynn RF, Bigger BW. Hematopoietic stem cell and gene therapy corrects primary neuropathology and behavior in mucopolysaccharidosis IIIA mice. Mol Ther. 2012 Aug;20(8):1610-21. doi: 10.1038/mt.2012.82. Epub 2012 May 1. PMID 22547151

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrolled 12 participants and 4 participants were included in each of the 3 dose groups.
Groups:
- HGT-1410 10 mg: HGT-1410/rhHNS 10 milligram (mg) monthly via an intrathecal drug delivery device (IDDD) (every 28 [±7 days]) for a total of 6 months.
- HGT-1410 45 mg: HGT-1410/rhHNS 45 mg monthly via an IDDD (every 28 [±7 days]) for a total of 6 months.
- HGT-1410 90 mg: HGT-1410/rhHNS 45 mg dose every 14 [±2 days] for a monthly total dose of 90 mg via an IDDD for 6 months.
Period: Overall Study
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HGT-1410 10 mg: HGT-1410/rhHNS 10 mg monthly via an IDDD (every 28 [±7 days]) for a total of 6 months.
- Total: Total of all reporting groups
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.15 (4.7) | 9.07 (9.8) | 10.64 (8.7) | 9.618 (7.2941)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 3 | 2 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Serious Adverse Events (SAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that did not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAEs) were defined as all adverse events (AEs) from the time of the surgery for IDDD implantation to the last follow up contact, 30 (±7) days after the end of study (EOS) procedures.
Time Frame: Baseline to week 30 (follow-up)
Population: Safety population was defined as all enrolled participants who received at least 1 dose (full or partial) of study drug.
Measure: Number; unit: events
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
events | 5 | 3 | 2

2. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAE)
Description: as for outcome 1
Time Frame: Baseline to week 30 (follow-up)
Population: Safety population.
Measure: Number; unit: events
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
events | 71 | 42 | 55

3. Primary Outcome: Summary of Anti-rhHNS Antibody Status in Cerebrospinal Fluid (CSF) by Recombinant Human Heparan N-Sulfatase (rhHNS) Dose Group
Description: Participants with positive, negative and missing status were reported.
Time Frame: Baseline, Week 26
Population: Intent to treat (ITT) population was defined as all enrolled participants who received at least 1 dose (full or partial) of study drug.
Measure: Number; unit: participants
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
participants
  Negative (Baseline) | 4 | 4 | 4
  Positive (Baseline) | 0 | 0 | 0
  Missing (Baseline) | 0 | 0 | 0
  Negative (Week 26) | 1 | 1 | 2
  Positive (Week 26) | 0 | 0 | 0
  Missing (Week 26) | 3 | 3 | 2

4. Primary Outcome: Summary of Anti-rhHNS Antibody Status in Serum by Recombinant Human Heparan N-Sulfatase (rhHNS) Dose Group
Description: Participants with positive, negative and missing status were reported.
Time Frame: Baseline, Week 26
Population: ITT population
Measure: Number; unit: participants
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
participants
  Negative (Baseline) | 4 | 3 | 3
  Positive (Baseline) | 0 | 1 | 1
  Missing (Baseline) | 0 | 0 | 0
  Negative (Week 26) | 1 | 2 | 2
  Positive (Week 26) | 2 | 0 | 0
  Missing (Week 26) | 1 | 2 | 2

5. Primary Outcome: Number of Participants With Intrathecal Drug Device (IDDD) Failures at Week 26
Description: Participants with IDDD failures were reported.
Time Frame: Week 26
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
participants | 3 | 2 | 1

6. Secondary Outcome: Change From Baseline in Developmental Quotient (DQ) Using Bayley Scales of Infant Development Third Edition (BSID III) and Kaufman Assessment Battery for Children Second Edition (KABC II) at Week 22
Description: BSID-III was used to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers. This measure consists of a series of developmental play tasks. Raw scores of successfully completed items are converted to scale scores and to composite scores. The mean composite score is 100 and the standard deviation (SD) is 15.Higher scores are indicative of decreased development. KABC-II was an individually administered measure of the processing and reasoning abilities of children and adolescents between the ages of 3 and 18 years and is an alternative to BSID-III. BSID-III DQ score was based on the Cognitive domain. The DQ score was calculated from the data obtained from either BSID-III/KABC-II mental age equivalent of the child in months divided by the calendar age in months (multiplied by 100 to give percentage points).
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  Baseline (n= 2, 4, 4) | 51.91 (27.292) | 43.24 (23.112) | 51.87 (36.095)
  Change at Week 22 (n= 2, 4, 4) | -13.6 (8.886) | -0.89 (4.341) | -4.91 (7.769)

7. Secondary Outcome: Change From Baseline in Four Point Scoring System/Total Disability Score (FPSS/TDS) at Week 22 and Week 26 (EOS)
Description: FPSS is a sanfilippo-specific disability assessment which assesses motor function, expressive/speech language, and cognitive function on a 0 to 3 point scale. A score of 3 points is assigned for normal function, 2 points for beginning of regression, 1 point for severe level of regression, and 0 points for lost skills. The total disability score (TDS) is the average (0-3) of the motor skills (MS), speech abilities (SA), and cognitive function (CF) scores. Lower scores indicate developmental regression.
Time Frame: Baseline, Week 22, Week 26
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  MS: Baseline (n= 4, 3, 4) | 2.5 (0.58) | 3 (0) | 3 (0)
  MS: Change at Week 22 (n= 4, 3, 4) | 0.3 (0.5) | 0 (0) | 0 (0)
  MS: Change at Week 26/EOS (n=2,2,3) | 0 (0) | 0 (0) | 0 (0)
  SA: Baseline (n= 4, 3, 4) | 2 (0.82) | 2 (0) | 2 (0.82)
  SA: Change at Week 22 (n= 4, 3, 4) | -0.5 (0.58) | 0.3 (0.58) | 0.3 (0.5)
  SA: Change at Week 26/EOS (n= 2, 2, 3) | -0.5 (0.71) | 0 (0) | 0.3 (0.58)
  CF: Baseline (n= 4, 3, 4) | 2.3 (0.5) | 0.5 (0.58) | 2.8 (0.5)
  CF: Change at Week 22 (n= 4, 3, 4) | 0 (0) | 0 (0) | 0 (0)
  CF: Change at Week 26/EOS (n= 2, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  TDS: Baseline (n= 4, 3, 4) | 2.25 (0.569) | 2.44 (0.192) | 2.58 (0.319)
  TDS: Change at Week 22 (n= 4, 3, 4) | -0.08 (0.319) | 0.11 (0.192) | 0.08 (0.167)
  TDS: Change at Week 26/EOS (n= 2, 2, 3) | -0.17 (0.236) | 0 (0) | 0.11 (0.192)

8. Secondary Outcome: Change From Baseline in Sanfilippo Behavioral Rating Scale (SBRS) at Week 22 and Week 26 (EOS)
Description: SBRS a parent-scored behavioral inventory measuring: comprehensive language skills, expressive language skills, tantrums, mood and emotions, and other behaviors not otherwise classified. Subscale items are scored 0=Never, 1=Occasionally(5-10%), 2=Sometimes (25%), 3=About half the time, 4=Often(75%), 5=Almost always (90%), 6=Always. Summary scores are the sum of responses within a given domain. Higher values = undesirable behavior. Total score range listed below with the abbreviations. Current Communication (CC)(0-42), Past Communication (PC)(0-42), Orality (0-36), Body Movements (BM)(0-30), Interaction With Objects (IWO)(0-24), Activity And Routines (AAR)(0-36), Emotional Function (EF)(0-18), Safety-consciousness (SC)(0-18), Fearfulness (0-36), Social Interaction (SI)(0-36), Eye Contact (EC)(0-18), Emotional Engagement (EE)(0-18), Comfort Seeking (CS)(0-30), Attention (0-18), Self-control/Compliance (SCC)(0-18), Mood, Anger/Aggression (MAA)(0-42), Self-gratification (SG)(0-24).
Time Frame: Baseline, Week 22, Week 26/EOS
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  CC: Baseline (n= 4, 4, 2) | 8.0 (5.48) | 6.3 (6.85) | 10.0 (5.66)
  CC: Change at Week 22 (n= 4, 4, 2) | 5.0 (13.44) | -0.3 (1.26) | 1.5 (2.12)
  CC: Change at Week 26/EOS (n= 3, 2, 2) | 1.3 (12.5) | -1.0 (1.41) | 1.5 (2.12)
  PC: Baseline (n= 3, 2, 4) | 7.3 (6.03) | 8.5 (12.02) | 11.0 (11.37)
  PC: Change at Week 22 (n= 1, 0, 1) | -8.0 (NA) — Not applicable (NA) signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  PC: Change at Week 26/EOS (n= 0, 0, 0) | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  Orality: Baseline (n= 2, 3, 3) | 7.0 (9.9) | 10.3 (2.08) | 17.3 (10.26)
  Orality: Change at Week 22 (n= 2, 3, 1) | 2.0 (2.83) | 6.0 (5.29) | 4.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  Orality: Change at Week 26/EOS (n= 1, 1, 1) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 5 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 4 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  BM: Baseline (n= 4, 4, 2) | 5.0 (4.55) | 2.5 (2.08) | 12.0 (2.83)
  BM: Change at Week 22 (n= 3, 4, 2) | 2.3 (3.51) | 2 (2.45) | -2.0 (2.83)
  BM: Change at Week 26/EOS (n= 3, 2, 2) | 0.3 (1.53) | 0 (0) | -2.0 (2.83)
  IWO: Baseline (n= 4, 3, 4) | 4.5 (3.11) | 10.3 (2.08) | 8.5 (7.9)
  IWO: Change at Week 22 (n= 4, 3, 3) | 3.3 (4.27) | -2.0 (4.58) | -2.0 (3.46)
  IWO: Change at Week 26/EOS (n= 2, 1, 3) | 1.0 (1.41) | -1.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -2.0 (3.46)
  AAR: Baseline (n= 1, 3, 4) | 6.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 14.3 (3.06) | 12.3 (9.46)
  AAR: Change at Week 22 (n= 1, 3, 4) | 8.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0.7 (0.58) | -1.3 (6.08)
  AAR: Change at Week 26/EOS (n= 0, 1, 3) | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 1.7 (2.08)
  EF: Baseline (n= 3, 4, 4) | 2.0 (3.46) | 2.5 (3.11) | 7.5 (5.0)
  EF: Change at Week 22 (n= 3, 4, 4) | 2.0 (3.46) | 2.5 (3.11) | 7.5 (5.0)
  EF: Change at Week 26/EOS (n= 2, 2, 3) | 5.0 (1.41) | 0.5 (0.71) | -1.31 (3.06)
  SC: Baseline (n= 4, 4, 4) | 7.8 (5.44) | 9.5 (1.91) | 11.5 (7.9)
  SC: Change at Week 22 (n= 4, 4, 4) | 0.5 (1.0) | 1.8 (5.74) | -0.8 (2.5)
  SC: Change at Week 26/EOS (n= 3, 2, 3) | -1.0 (2.65) | -3.0 (2.83) | -1.0 (3.0)
  Fearfulness: Baseline (n= 3, 3, 3) | 7.0 (7.81) | 10.3 (8.74) | 11.0 (6.08)
  Fearfulness: Change at Week 22 (n= 3, 3, 3) | 2.7 (1.15) | -1.0 (5.2) | 2.0 (1.73)
  Fearfulness: Change at Week 26/EOS (n= 2, 1, 3) | 2.5 (2.12) | -5 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 2.3 (1.53)
  SI: Baseline (n= 4, 4, 4) | 11.0 (3.37) | 12.5 (2.38) | 14.5 (6.76)
  SI: Change at Week 22 (n= 4, 3, 4) | 3.0 (4.76) | 0.3 (4.04) | -0.5 (3.7)
  SI: Change at Week 26/EOS (n= 3, 2, 3) | 0 (8.0) | -3.5 (4.95) | -0.7 (4.62)
  EC: Baseline (n= 4, 4, 3) | 2.8 (3.59) | 5.5 (3.7) | 6.7 (5.77)
  EC: Change at Week 22 (n= 4, 4, 3) | 1.5 (1.73) | 0 (3.27) | -1.0 (2.65)
  EC: Change at Week 26/EOS (n= 3, 2, 3) | 0.3 (0.58) | -2.0 (2.83) | -0.7 (3.06)
  EE: Baseline (n= 2, 4, 4) | 8.5 (4.95) | 7.3 (1.71) | 8.3 (3.3)
  EE: Change at Week 22 (n= 1, 4, 4) | 2.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -0.5 (1.29) | -0.8 (2.87)
  EE: Change at Week 26/EOS (n= 0, 2, 3) | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -1.0 (1.41) | 0.7 (1.15)
  CS: Baseline (n= 4, 3, 4) | 10.3 (5.32) | 10.3 (3.06) | 16.5 (6.56)
  CS: Change at Week 22 (n= 3, 3, 3) | 1.7 (4.73) | -1.7 (3.06) | -2.3 (3.21)
  CS: Change at Week 26/EOS (n= 2, 1, 3) | 0 (1.41) | -1.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -2.3 (3.21)
  Attention: Baseline (n= 4, 4, 4) | 8.3 (4.65) | 8.8 (1.26) | 10.5 (7.72)
  Attention: Change at Week 22 (n= 4, 4, 4) | 1.0 (3.16) | 2.5 (2.38) | 2.3 (1.71)
  Attention: Change at Week 26/EOS (n= 2, 2, 3) | 1.5 (2.12) | 0.5 (0.71) | 3.3 (1.15)
  SCC: Baseline (n= 4, 4, 4) | 8.0 (4.97) | 7.3 (2.22) | 10.0 (7.3)
  SCC: Change at Week 22 (n= 3, 4, 4) | 0.3 (4.51) | 3.3 (3.2) | 2.0 (1.83)
  SCC: Change at Week 26/EOS (n= 3, 2, 3) | 0.7 (4.04) | 0.5 (0.71) | 2.7 (1.53)
  MAA: Baseline (n= 4, 3, 4) | 5.3 (4.11) | 9.7 (3.51) | 17.3 (15.65)
  MAA: Change at Week 22 (n= 2, 3, 4) | 5.5 (7.78) | 3.3 (5.13) | -0.3 (2.5)
  MAA: Change at Week 26/EOS (n= 3, 1, 3) | 1.7 (3.06) | 4.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -0.7 (2.89)
  SG: Baseline (n= 4, 3, 4) | 0.5 (1.0) | 0.3 (0.58) | 4.5 (5.26)
  SG: Change at Week 22 (n= 3, 3, 4) | -0.7 (1.15) | 2.0 (1.0) | -1.0 (4.08)
  SG: Change at Week 26/EOS (n= 3, 1, 3) | 0.3 (0.58) | 1.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 1.0 (1.0)

9. Secondary Outcome: Change From Baseline in Developmental Quotient (DQ) Using Vineland Adaptive Behavioral Scales Second Edition (VABS-II) at Week 22
Description: VABS-II measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. It is an instrument that supports the diagnosis of intellectual and developmental disabilities in participants. This test measures 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other four domains). Scoring is 'Usually' = 2, 'Sometimes'/Partially' = 1 or 'Never' = 0. The raw scores will be converted to domain standard scores (mean 100, SD 15). Higher scores indicate undesirable behavior. The Overall DQ score was calculated from the mean age-equivalent score obtained by averaging out the age equivalent scores for all the sub-domains except for Gross and Fine motor skills.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  Baseline (n= 4, 4, 4) | 44.78 (24.747) | 47.24 (26.612) | 47.71 (33.687)
  Change at Week 22 (n= 2, 2, 2) | -11.38 (12.478) | -23.96 (10.014) | -10.18 (13.333)

10. Secondary Outcome: Change From Baseline in Movement Assessment Battery for Children Second Edition (MABC-2) at Week 26 (EOS)
Description: Movement Assessment Battery for Children, Second Edition (MABC-II) was to be used to identify, describe and guide the treatment of motor impairment in children from 3.0 to 16:11 years of age. As per statistical analysis plan, the outcome was to be assessed only if greater than (>) 50 percent (%) of participants were available for the evaluation.
Time Frame: Baseline, Week 26/EOS
Population: This outcome measure was not analyzed as it does not meet the pre-specified SAP criteria (outcome was to be assessed only if greater than (>) 50 percent (%) of participants were available for the evaluation).
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Using Child Health Questionnaire™ Parent Form 50 (CHQ-PF50) Questions at Week 22 and Week 26 (EOS)
Description: CHQ-PF50 which was designed to measure the physical and psychosocial well-being of children 5 years to 18 years of age, consists of 13 health concepts including 11 multi-item and 2 single item scales: Physical Function (PF), Role/Social-Emotional/Behavioral (REB), Role/Social-Physical (RP), bodily pain (BP), General Behavior (BE), Mental Health (MH), Self Esteem (SE), General Health Perceptions (GH), Change in Health (CH), Parental Impact-Emotional (PE), Parental Impact-Time (PT), Family Activities (FA), and Family Cohesion (FC). Transformed scores for all subscales range from 0 to 100, with a higher score indicating better health. Physical and Psychosocial Summary measures (SM) were scored with the use of norm-based methods that standardize the scores to a mean (± Standard Deviation) of 50 ± 10 on the basis of an assessment of the general United States population. Higher values represent better health.
Time Frame: Baseline, Week 22, Week 26/EOS
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  PF: Baseline (n= 2, 4, 2) | 66.67 (47.14) | 80.28 (35.141) | 66.67 (23.57)
  PF: Change at Week 22 (n= 2, 4, 2) | -8.33 (51.069) | -16.39 (23.047) | 5.56 (15.713)
  PF: Change at Week 26/EOS (n= 1, 2, 1) | 33.33 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -24.44 (34.57) | -11.11 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  RP: Baseline (n= 2, 4, 2) | 66.67 (47.14) | 50 (57.735) | 66.67 (47.14)
  RP: Change at Week 22 (n= 2, 4, 2) | 8.33 (11.785) | 8.33 (16.667) | 0 (0)
  RP: Change at Week 26/EOS (n= 1, 2, 1) | 33.33 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  BP: Baseline (n= 2, 4, 2) | 90 (14.14) | 67.5 (29.86) | 30 (0)
  BP: Change at Week 22 (n= 2, 4, 2) | -20 (56.57) | 7.5 (15) | 45 (7.07)
  BP: Change at Week 26/EOS (n= 1, 2, 1) | 20 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (0) | 50 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  GH: Baseline (n= 2, 4, 2) | 45.42 (2.946) | 27.92 (21.457) | 33.33 (23.57)
  GH: Change at Week 22 (n= 2, 4, 2) | -7.75 (38.537) | -5.21 (10.417) | 11.25 (15.91)
  GH: Change at Week 26/EOS(n= 1, 2, 1) | 17.5 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (0) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  REB: Baseline (n= 2, 4, 2) | 66.67 (47.14) | 41.67 (50) | 50 (70.711)
  REB: Change at Week 22 (n= 2, 4, 2) | -38.89 (86.424) | 11.11 (64.788) | 0 (0)
  REB: Change at Week 26/EOS (n= 1, 2, 1) | 22.22 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (0) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  BE: Baseline (n= 2, 4, 2) | 62.5 (17.678) | 61.04 (15.296) | 45.83 (11.785)
  BE: Change at Week 22 (n= 2, 4, 2) | 12.08 (8.839) | -2.92 (15.716) | -2.08 (2.946)
  BE: Change at Week 26/EOS (n= 1, 2, 1) | 30.83 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -14.37 (14.437) | -8.33 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  MH: Baseline (n= 2, 4, 2) | 75 (7.07) | 68.8 (10.31) | 10 (14.14)
  MH: Change at Week 22 (n= 2, 4, 2) | 0 (21.21) | -2.5 (16.58) | 17.5 (17.68)
  MH: Change at Week 26/EOS (n= 1, 2, 1) | 15 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -5 (7.07) | 5 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  SE: Baseline (n= 2, 4, 2) | 62.5 (5.893) | 61.46 (18.122) | 47.92 (14.731)
  SE: Change at Week 22 (n= 2, 4, 2) | 0 (11.785) | -3.13 (7.116) | -4.17 (5.893)
  SE: Change at Week 26/EOS (n= 1, 2, 1) | 16.67 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 8.33 (11.785) | -8.33 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  PE: Baseline (n= 2, 4, 2) | 66.67 (47.14) | 27.08 (22.948) | 20.83 (17.678)
  PE: Change at Week 22 (n= 2, 4, 2) | -8.33 (82.496) | -2.08 (14.232) | 4.17 (5.893)
  PE: Change at Week 26/EOS (n= 1, 2, 1) | 16.67 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -4.17 (5.893) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  PT: Baseline (n= 2, 4, 2) | 50 (70.711) | 33.33 (28.689) | 5.56 (7.857)
  PT: Change at Week 22 (n= 2, 4, 2) | 11.11 (62.854) | -5.56 (26.45) | 16.67 (23.57)
  PT: Change at Week 26/EOS (n= 1, 2, 1) | 44.44 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -5.56 (23.57) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  FA: Baseline (n= 2, 4, 2) | 56.25 (61.872) | 42.71 (13.767) | 10.42 (14.731)
  FA: Change at Week 22 (n= 2, 4, 2) | 0 (58.926) | -7.29 (13.767) | 0 (0)
  FA: Change at Week 26/EOS (n= 1, 2, 1) | 16.67 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -6.25 (2.946) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  FC: Baseline (n= 2, 4, 2) | 57.5 (38.89) | 72.5 (14.43) | 15.0 (21.21)
  FC: Change at Week 22 (n= 2, 4, 2) | 27.5 (38.89) | -6.3 (12.5) | 15.0 (21.21)
  FC: Change at Week 26/EOS (n= 1, 2, 1) | 55.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | 0 (0) | 30 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  SM Physical: Baseline (n= 2, 4, 2) | 38.44 (23.545) | 31.62 (23.071) | 31.27 (18.193)
  SM Physical: Change at Week 22 (n= 2, 4, 2) | -4.63 (29.276) | -1.82 (6.112) | 9.21 (5.095)
  SM Physical: Change at Week 26/EOS (n= 1, 2, 1) | 17.25 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -4.99 (8.195) | 4.96 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure
  SM Psychosocial: Baseline (n= 2, 4, 2) | 42.16 (14.06) | 33.8 (10.879) | 17.57 (2.418)
  SM Psychosocial: Change at Week 22 (n= 2, 4, 2) | -1.18 (23.341) | -0.26 (14.004) | 2.27 (4.972)
  SM Psychosocial:Change at Week 26/EOS (n= 1, 2, 1) | 13.64 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure | -1.58 (2.584) | -2.29 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure

12. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Using Infant Toddler Quality of Life Questionnaire™ (ITQOL) at Week 22 and Week 26 (EOS)
Description: ITQOL is a generic, validated health status measure for children aged 2 months up to 5 years, including items and scales to measure aspects of physical functioning, development, pain, mood, behavior, general health and impact on parents. The ITQOL consists of 97 items that are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health). The score range for all individual subscales is 0 (worst health) to 100 (best health). Abbreviation: Overall Health (OH), Physical Abilities (PA), Growth And Development (GAD), Bodily Pain (BP), Temperament And Moods (TAM), General Behavior (GEB), Global Behavior (GLB), Getting Along (GA), General Health Perceptions (GHP), PI-Emotion (PIE), PI-Time (PIT), Family Cohesion (FC).
Time Frame: Baseline, Week 22, Week 26/EOS
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  OH: Baseline (n= 2, 3, 2) | 80 (28.28) | 56.7 (49.07) | 65 (49.5)
  OH: Change at Week 22 (n= 2, 2, 2) | 0 (0) | -12.5 (17.68) | 15 (21.21)
  OH: Change at Week 26/EOS (n= 1, 0, 0) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  PA: Baseline (n= 2, 3, 2) | 83.35 (9.405) | 75.57 (39.496) | 93.35 (4.738)
  PA: Change at Week 22 (n= 2, 2, 2) | 5 (11.738) | 1.65 (11.809) | -1.7 (2.404)
  PA: Change at Week 26/EOS (n= 1, 0, 0) | -3.3 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  GAD: Baseline (n= 2, 3, 2) | 57.2 (18.102) | 60.83 (25.658) | 56.8 (6.081)
  GAD: Change at Week 22 (n= 2, 2, 2) | -14.7 (28.709) | -22.5 (7.071) | 18.2 (0.99)
  GAD: Change at Week 26/EOS (n= 1, 0, 0) | 3.1 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  BP: Baseline (n= 2, 3, 2) | 95.85 (5.869) | 58.33 (36.294) | 62.5 (29.416)
  BP: Change at Week 22 (n= 2, 2, 2) | -29.2 (17.678) | 25 (11.738) | 12.5 (41.154)
  BP: Change at Week 26/EOS (n= 1, 0, 0) | -16.7 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  TAM: Baseline (n= 2, 3, 2) | 72.2 (17.678) | 68.97 (21.731) | 52.8 (15.698)
  TAM: Change at Week 22 (n= 2, 2, 2) | -23.6 (21.637) | -2.75 (33.446) | -5.6 (19.658)
  TAM: Change at Week 26/EOS (n= 1, 0, 0) | -12.8 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  GEB: Baseline (n= 2, 3, 2) | 58.35 (32.456) | 34.73 (17.465) | 12.5 (5.94)
  GEB: Change at Week 22 (n= 2, 2, 2) | -12.5 (8.91) | 7.25 (25.102) | 18.75 (0.071)
  GEB: Change at Week 26/EOS (n= 1, 0, 0) | -8.3 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  GLB: Baseline (n= 2, 3, 2) | 57.5 (38.89) | 40 (34.64) | 0 (0)
  GLB: Change at Week 22 (n= 2, 2, 2) | -15 (21.21) | 0 (42.43) | 0 (0)
  GLB: Change at Week 26/EOS (n= 1, 0, 0) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  GA: Baseline (n= 2, 3, 2) | 62.5 (17.678) | 55 (15) | 35.85 (1.202)
  GA: Change at Week 22 (n= 2, 2, 2) | -22.5 (10.607) | -2.5 (22.345) | -1.65 (16.476)
  GA: Change at Week 26/EOS (n= 1, 0, 0) | -16.7 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  GHP: Baseline (n= 2, 3, 2) | 48.9 (4.808) | 31.8 (20.178) | 57.95 (36.982)
  GHP: Change at Week 22 (n= 2, 2, 2) | -18.2 (22.486) | -5.7 (1.556) | -3.8 (11.879)
  GHP: Change at Week 26/EOS (n= 1, 0, 0) | 0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  PIE: Baseline (n= 2, 3, 2) | 78.55 (30.335) | 48.83 (33.024) | 41.65 (23.547)
  PIE: Change at Week 22 (n= 2, 2, 2) | -35.7 (25.314) | -3.6 (25.314) | 4.75 (3.323)
  PIE: Change at Week 26/EOS (n= 1, 0, 0) | -17.8 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  PIT: Baseline (n= 2, 3, 2) | 73.8 (37.052) | 49.2 (26.264) | 45.25 (63.993)
  PIT: Change at Week 22 (n= 2, 2, 2) | -33.35 (6.718) | 7.2 (23.617) | 23.8 (20.223)
  PIT: Change at Week 26/EOS (n= 1, 0, 0) | -28.6 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  FC: Baseline (n= 2, 3, 2) | 85 (0) | 76.7 (14.43) | 42.5 (60.1)
  FC: Change at Week 22 (n= 2, 2, 2) | -12.5 (17.68) | -12.5 (17.68) | -27.5 (38.89)
  FC: Change at Week 26/EOS (n= 1, 0, 0) | -25 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | NA (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.

13. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Using Child Health Questionnaire™ Child Form 87 (CHQ-CF87) at Week 26 (EOS)
Description: CHQ-CF87 form was designed to be a self-report for participants 10 years and older. It consists of 87 questions and contains the same scales as the PF-50, (with the omission of the parental impact scales and there are no psychosocial and physical summary scores derived). As per statistical analysis plan, the outcome was to be assessed only if greater than (>) 50 percent (%) of participants were available for the evaluation.
Time Frame: Baseline, Week 26/EOS
Population: as for outcome 10
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Using Children's Sleep Habits Rating Scale at Week 22 and Week 26 (EOS)
Description: Children's sleep habits rating scale consisting of 35 item parent questionnaire sleep screening tool. Items are scored on a 3-point scale from 1 (rarely) to 3 (usually) with a Total Sleep Disturbance score (TSDS) ranging from 35-105. Eight subscale scores are totaled to create the TSDS. The subscales are: Bedtime Resistance (BR)(6 items, score = 6-18), Sleep Duration (SD)(3 items, score = 3-9), Parasomnias (P)(7 items, score = 7-21), Sleep Disordered Breathing (SDB)(3 items, score = 3-9), Night Waking (NW)(3 items, score = 3-9), Daytime Sleepiness (DS)(8 items, score = 8-24), Sleep Anxiety (SA)(4 items, score = 4-12), and Sleep Onset Delay (SOD)(1 item, score = 1-3). The questionnaire was designed for children aged 4 through 12 years. A higher score is indicative of more disturbed sleep.
Time Frame: Baseline, Week 22, Week 26/EOS
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
units on a scale
  BR: Baseline (n= 4, 4, 4) | 8.8 (1.89) | 7.3 (2.5) | 11.5 (4.65)
  BR: Change at Week 22 (n= 4, 4, 4) | -1.3 (1.89) | 1.3 (0.96) | -0.8 (0.96)
  BR: Change at Week 26/EOS (n= 3, 2, 2) | -1 (1) | 1 (1.41) | 0 (0)
  SOD: Baseline (n= 4, 4, 4) | 1.5 (1) | 1.8 (0.96) | 2.3 (0.96)
  SOD: Change at Week 22 (n= 4, 4, 4) | 0 (0.82) | 0 (0.82) | 0 (0.82)
  SOD: Change at Week 26/EOS (n= 3, 2, 2) | -0.3 (0.58) | -0.5 (0.71) | 0 (1.41)
  SD: Baseline (n= 4, 4, 4) | 5.3 (2.22) | 6.5 (2.65) | 6 (2.16)
  SD: Change at Week 22 (n= 4, 4, 4) | -0.8 (2.99) | -0.5 (1.29) | 1.3 (1.5)
  SD: Change at Week 26/EOS (n= 3, 2, 2) | -1.7 (2.89) | -1 (1.41) | 1 (1.41)
  SA: Baseline (n= 4, 4, 4) | 7 (1.15) | 6 (1.41) | 8.3 (3.3)
  SA: Change at Week 22 (n= 4, 4, 3) | -1.5 (1.91) | 0.8 (1.71) | -0.3 (0.58)
  SA: Change at Week 26/EOS (n= 3, 2, 2) | -0.7 (1.15) | 0 (1.41) | -0.5 (0.71)
  NW: Baseline (n= 4, 4, 4) | 4.3 (1.5) | 5.5 (1.91) | 5.8 (2.5)
  NW: Change at Week 22 (n= 4, 4, 4) | -0.3 (2.06) | 0 (1.63) | -0.5 (0.58)
  NW: Change at Week 26/EOS (n= 3, 2, 2) | -1 (1.73) | -0.5 (0.71) | 0 (0)
  P: Baseline (n= 2, 4, 4) | 8.5 (0.71) | 10 (2.31) | 12 (2.94)
  P: Change at Week 22 (n= 2, 4, 4) | -1 (0) | 0.3 (3.4) | -0.3 (2.87)
  P: Change at Week 26/EOS (n= 1, 2, 2) | -1 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -1 (0) | -0.5 (0.71)
  SDB: Baseline (n= 4, 4, 4) | 3.3 (0.5) | 4.3 (0.5) | 5.8 (3.2)
  SDB: Change at Week 22 (n= 4, 4, 3) | 0.8 (0.96) | 0.5 (1.73) | -1.7 (2.89)
  SDB: Change at Week 26/EOS(n= 3, 2, 2) | 0.7 (1.15) | -0.5 (0.71) | 0 (0)
  DS: Baseline (n= 4, 4, 4) | 9.5 (1.29) | 11.5 (3.87) | 11.3 (3.4)
  DS: Change at Week 22 (n= 4, 4, 4) | -0.3 (0.5) | 0.5 (0.58) | 0.5 (2.65)
  DS: Change at Week 26/EOS (n= 3, 2, 2) | 0.7 (1.15) | 1 (0) | 1 (1.41)
  TSDS: Baseline (n= 2, 4, 4) | 42.5 (2.12) | 50.3 (12.28) | 58.8 (16.82)
  TSDS: Change at Week 22 (n= 2, 4, 2) | 1.5 (4.95) | 2 (5.83) | 2 (5.66)
  TSDS: Change at Week 26/EOS (n= 1, 2, 2) | -2 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -2 (4.24) | 1 (2.83)

15. Secondary Outcome: Number of Participants With Accumulation of Recombinant Human Heparan N-Sulfatase (rhHNS) in Cerebrospinal Fluid (CSF) at Week 22
Description: Cerebrospinal fluid samples were collected from participants through an implanted IDDD or via lumbar puncture (LP) immediately prior to each administration of HGT-1410.
Time Frame: Baseline, Week 22
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
participants | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Concentration of Heparan Sulfate and Heparan Sulfate Derivatives in Cerebrospinal Fluid (CSF) at Week 6, 10, 14, 18, 22 and 26(EOS)
Description: Levels of heparan sulfate and its derivatives were evaluated using the proprietary Sensi-Pro (SP) high-performance liquid chromatography (HPLC) based assay. Abbreviation: SP Total Heparan Sulfate (SPTHS), SP Non-Reducing End Assay (SPNREA),
Time Frame: Baseline, Week 6, 10, 14, 18, 22 and 26(EOS)
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: picomole per milliliter (pmol/mL)
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
picomole per milliliter (pmol/mL)
  SPTHS: Baseline (n= 4, 4, 4) | 90570.5 (38088.67) | 69049.7 (42659.28) | 83287.0 (26012.16)
  SPTHS: Change at Week 6 (n= 4, 2, 2) | -34167.7 (20439.34) | -41331.4 (38967.66) | -65862.6 (23010.52)
  SPTHS: Week 10 (n= 4, 4, 3) | -41825.4 (13482.5) | -39441.8 (29771.14) | -54343.7 (25891.78)
  SPTHS: Change at Week 14 (n= 4, 3, 3) | -40309 (15107.94) | -32249.2 (21862.89) | -64763.9 (25285.97)
  SPTHS: Change at Week 22 (n= 4, 4, 4) | -35469.5 (20922.54) | -44669.5 (38360.07) | -60931.7 (20699.36)
  SPNREA: Baseline (n= 4, 4, 4) | 1255.93 (471.403) | 1198.34 (627.436) | 1487.67 (329.790)
  SPNREA: Change at Week 6 (n= 4, 2, 2) | -213.25 (330.836) | -677.79 (393.281) | -1022.53 (163.905)
  SPNREA: Change at Week 10 (n= 4, 4, 3) | -411.77 (268.961) | -533.38 (476.259) | -788.65 (390.761)
  SPNREA: Change at Week 14 (n= 4, 3, 3) | -359.15 (272.695) | -491.24 (177.701) | -1033.58 (371.566)
  SPNREA: Change at Week 22 (n= 4, 4, 4) | -254.07 (333.649) | -686.13 (517.558) | -877.84 (435.044)

17. Secondary Outcome: Change From Baseline in Brain Magnetic Resonance Imaging (MRI) at Week 22
Description: Brain MRI was measured for grey matter volume (GMV) , white matter volume (WMV) and Intracranial cerebrospinal fluid Volume (ICSFV) (Ventricles + Additional CSF Space).
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
milliliter (mL)
  GMV: Baseline | 550.5 (111.043) | 534.25 (117.291) | 600.28 (67.884)
  GMV: Change at Week 22 | -42.84 (36.793) | -33.7 (24.161) | -32.87 (36.862)
  WMV: Baseline | 403.72 (105.575) | 348.28 (76.854) | 442.45 (79.814)
  WMV: Change at Week 22 | -2.86 (13.997) | 3.33 (11.419) | -0.44 (9.793)
  ICSFV: Baseline | 26.152 (9.2975) | 22.904 (20.8459) | 20.925 (15.9681)
  ICSFV: Change at Week 22 | 4.739 (4.6455) | 2.886 (3.9153) | 7.375 (6.6573)

18. Secondary Outcome: Change From Baseline in Mean Auditory Brainstem Response (ABR) at Week 22
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Mean ABR air and bone conduction threshold were assessed. Mean ABR bone conduction threshold was not possible to be reported as there was insufficient data to be analysed.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Decibel Above Normal Adult Hearing Level
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
Decibel Above Normal Adult Hearing Level
  Right Ear: Baseline (n= 1, 2, 3) | 62.5 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | 56.25 (8.839) | 49.17 (14.216)
  Right Ear: Change at Week 22 (n= 1, 2, 3) | -10.0 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -3.75 (15.91) | -0.83 (22.407)
  Left Ear: Baseline (n= 2, 2, 4) | 52.5 (10.607) | 55.0 (7.071) | 44.38 (24.696)
  Left Ear: Change at Week 22 (n= 2, 2, 4) | 5.0 (7.071) | -5.0 (14.142) | 3.13 (10.68)

19. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Latencies
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. The Inter-peak Latencies (IPL) were calculated by subtracting the absolute latencies (AL). The Inter-aural Latencies (IAL) were calculated by subtracting the absolute wave V latencies of the right and left ear. IAL, IPL and AL were reported. Abbreviation: Right Ear (RE), Left Ear (LE), Wave (W), Wave V (WV)
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
millisecond (ms)
  RE,IPL I-III: Baseline (n= 3, 3, 3) | 2.29 (0.257) | 2.53 (0.153) | 2.33 (0.193)
  RE,IPL I-III: Change at Week 22 (n= 3, 3, 2) | -0.09 (0.147) | -0.11 (0.183) | 0.07 (0.014)
  RE,IPL III-V: Baseline (n= 3, 3, 3) | 2.04 (0.24) | 2.17 (0.261) | 1.96 (0.119)
  RE,IPL III-V: Change at Week 22 (n= 3, 3, 2) | -0.08 (0.185) | -0.06 (0.304) | 0.06 (0.085)
  RE,IPL I-V: Baseline (n= 3, 3, 3) | 4.34 (0.047) | 4.71 (0.352) | 4.29 (0.238)
  RE,IPL I-V: Change at Week 22 (n= 3, 3, 3) | -0.17 (0.269) | -0.17 (0.187) | 0.2 (0.131)
  LE,IPL I-III: Baseline (n= 3, 3, 4) | 2.32 (0.206) | 2.53 (0.153) | 2.4 (0.303)
  LE,IPL I-III: Change at Week 22 (n= 3, 3, 3) | -0.01 (0.129) | -0.24 (0.065) | 0.11 (0.219)
  LE,IPL III-V: Baseline (n= 3, 3, 4) | 2.06 (0.255) | 2.15 (0.225) | 2.09 (0.311)
  LE,IPL III-V: Change at Week 22 (n= 3, 3, 3) | -0.02 (0.075) | 0.09 (0.091) | 0.06 (0.04)
  LE,IPL I-V: Baseline (n= 3, 3, 4) | 4.39 (0.264) | 4.68 (0.33) | 4.48 (0.394)
  LE,IPL I-V: Week 22 (n= 3, 3, 3) | -0.03 (0.185) | -0.15 (0.07) | 0.17 (0.191)
  IAL: Baseline (n= 3, 3, 3) | -0.05 (0.061) | -0.07 (0.058) | 0.07 (0.081)
  IAL: Change at Week 22 (n= 3, 3, 3) | 0.04 (0.301) | 0.28 (0.312) | 0.46 (0.849)
  AL-RE,WI: Baseline (n= 3, 3, 3) | 1.73 (0.237) | 1.59 (0.156) | 1.76 (0.012)
  AL-RE,WI: Change at Week 22 (n= 3, 3, 3) | 0 (0.466) | 0.46 (0.54) | 0.47 (0.987)
  AL-RE,WIII: Baseline (n= 3, 3, 2) | 4.02 (0.45) | 4.12 (0.197) | 4.09 (0.181)
  AL-RE,WIII: Change at Week 22 (n= 3, 3, 2) | -0.09 (0.355) | 0.35 (0.687) | -0.03 (0.042)
  AL-RE,WV: Baseline (n= 3, 3, 3) | 6.06 (0.283) | 6.3 (0.454) | 6.06 (0.227)
  AL-RE,WV: Change at Week 22 (n= 3, 3, 3) | -0.17 (0.478) | 0.29 (0.633) | 0.67 (1.109)
  AL-LE,WI: Baseline (n= 3, 3, 4) | 1.73 (0.13) | 1.68 (0.144) | 1.78 (0.233)
  AL-LE,WI: Change at Week 22 (n= 3, 3, 3) | -0.18 (0.111) | 0.16 (0.33) | 0.04 (0.16)
  AL-LE,WIII: Baseline (n= 3, 3, 4) | 4.05 (0.323) | 4.22 (0.189) | 4.18 (0.504)
  AL-LE,WIII: Change at Week 22 (n= 3, 3, 3) | -0.19 (0.165) | -0.08 (0.266) | 0.15 (0.306)
  AL-LE,WV: Baseline (n= 3, 3, 4) | 6.12 (0.278) | 6.36 (0.412) | 6.26 (0.612)
  AL-LE,WV: Change at Week 22 (n= 3, 3, 4) | -0.21 (0.178) | 0.01 (0.324) | 0.24 (0.227)

20. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Amplitudes
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR amplitudes by left ear (LE) and right ear (RE) were reported.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: microvolt (mcV)
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
microvolt (mcV)
  RE, Wave I: Baseline (n= 2, 3, 3) | 0.49 (0.042) | 0.42 (0.118) | 0.26 (0.097)
  RE, Wave I: Change at Week 22 (n= 2, 3, 3) | -0.23 (0.042) | -0.17 (0.147) | -0.03 (0.216)
  RE, Wave III: Baseline (n= 2, 3, 3) | 0.33 (0.156) | 0.35 (0.195) | 0.24 (0.113)
  RE, Wave III: Change at Week 22 (n= 2, 3, 2) | -0.05 (0.099) | -0.12 (0.117) | -0.16 (0.156)
  RE, Wave V: Baseline (n= 2, 3, 3) | 0.64 (0.403) | 0.47 (0.144) | 0.32 (0.101)
  RE, Wave V: Change at Week 22 (n= 2, 3, 3) | -0.28 (0.354) | -0.09 (0.145) | -0.14 (0.201)
  LE, Wave I: Baseline (n= 2, 3, 4) | 0.4 (0.028) | 0.44 (0.199) | 0.26 (0.133)
  LE, Wave I: Change at Week 22 (n= 2, 3, 3) | -0.1 (0.17) | 0.02 (0.221) | -0.01 (0.135)
  LE, Wave III: Baseline (n= 2, 3, 4) | 0.22 (0.106) | 0.38 (0.194) | 0.21 (0.102)
  LE, Wave III: Change at Week 22 (n= 2, 3, 3) | 0.05 (0.057) | -0.09 (0.188) | 0.02 (0.047)
  LE, Wave V: Baseline (n= 2, 3, 4) | 0.52 (0.269) | 0.48 (0.123) | 0.29 (0.17)
  LE, Wave V: Change at Week 22 (n= 2, 3, 4) | -0.13 (0.24) | -0.02 (0.134) | -0.01 (0.085)

21. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Amplitude Ratio
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR amplitudes(A), log-transformed amplitudes (LTA), square-root transformed amplitudes (STA) by left ear (LE) and right ear (RE) wave V/I in ratio was reported.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
ratio
  A-RE, Wave V/I: Baseline (n= 2, 2, 2) | 1.34 (0.94) | 1.09 (0.057) | 1.83 (0.403)
  A-RE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.14 (0.269) | 0.42 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -1.48 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  A-LE, Wave V/I: Baseline (n= 2, 2, 2) | 1.33 (0.764) | 1.26 (0.014) | 2.43 (2.341)
  A-LE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.37 (0.453) | 0.28 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -0.15 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  LTA-RE, Wave V/I: Baseline (n= 2, 2, 2) | 0.146 (0.7733) | 0.086 (0.0519) | 0.589 (0.2227)
  LTA-RE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.188 (0.3011) | 0.336 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -3.245 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  LTA-LE, Wave V/I: Baseline (n= 2, 2, 2) | 0.195 (0.6093) | 0.231 (0.0112) | 0.572 (1.1791)
  LTA-LE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.188 (0.1787) | 0.202 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -0.217 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  STA-RE, Wave V/I: Baseline (n= 2, 2, 2) | 1.116 (0.4212) | 1.044 (0.0271) | 1.347 (0.1496)
  STA-RE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.082 (0.1409) | 0.188 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -0.996 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.
  STA-LE, Wave V/I: Baseline (n= 2, 2, 2) | 1.128 (0.3385) | 1.122 (0.0063) | 1.449 (0.8078)
  STA-LE, Wave V/I: Change at Week 22 (n= 2, 1, 1) | 0.13 (0.1448) | 0.119 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure. | -0.09 (NA) — NA signifies standard deviation not reported as there was only 1 evaluable participant and data was not available for the specific measure.

22. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Log Transformed Latencies
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR log-transformed latencies (LTL) by left and right ear were reported.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: log transformed (latency [ms])
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
log transformed (latency [ms])
  LTL-RE, Wave I: Baseline (n= 3, 3, 3) | 0.54 (0.1326) | 0.461 (0.0956) | 0.567 (0.0066)
  LTL-RE, Wave I: Change at Week 22 (n= 3, 3, 3) | -0.006 (0.2585) | 0.242 (0.2791) | 0.179 (0.4104)
  LTL-RE, Wave III: Baseline (n= 3, 3, 3) | 1.387 (0.1121) | 1.416 (0.0483) | 1.409 (0.0439)
  LTL-RE, Wave III: Change at Week 22 (n= 3, 3, 2) | -0.019 (0.0882) | 0.074 (0.148) | -0.008 (0.0108)
  LTL-RE, Wave V: Baseline (n= 3, 3, 3) | 1.802 (0.0461) | 1.838 (0.0731) | 1.801 (0.0374)
  LTL-RE, Wave V: Change at Week 22 (n= 3, 3, 3) | -0.028 (0.0794) | 0.044 (0.0963) | 0.093 (0.1529)
  LTL-LE, Wave I: Baseline (n= 3, 3, 4) | 0.546 (0.0769) | 0.518 (0.0838) | 0.57 (0.1268)
  LTL-LE, Wave I: Change at Week 22 (n= 3, 3, 3) | -0.106 (0.0653) | 0.088 (0.1812) | 0.019 (0.0927)
  LTL-LE, Wave III: Baseline (n= 3, 3, 4) | 1.397 (0.0804) | 1.438 (0.0455) | 1.424 (0.1213)
  LTL-LE, Wave III: Change at Week 22 (n= 3, 3, 3) | -0.046 (0.0394) | -0.02 (0.0624) | 0.032 (0.0657)
  LTL-LE, Wave V: Baseline (n= 3, 3, 4) | 1.81 (0.045) | 1.849 (0.0658) | 1.831 (0.0955)
  LTL-LE, Wave V: Change at Week 22 (n= 3, 3, 4) | -0.034 (0.0281) | 0.002 (0.0494) | 0.036 (0.0338)

23. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Log Transformed Amplitude
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR log-transformed amplitudes (LTA) by left and right ear were reported.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: log transformed (amplitude [mcV])
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
log transformed (amplitude [mcV])
  LTA-RE, Wave I: Baseline (n= 2, 3, 3) | -0.715 (0.0867) | -0.893 (0.2741) | -1.379 (0.3627)
  LTA-RE, Wave I: Change at Week 22 (n= 2, 3, 3) | -0.659 (0.2456) | -0.76 (0.8475) | -0.24 (1.018)
  LTA-RE, Wave III: Baseline (n= 2, 3, 3) | -1.168 (0.4901) | -1.17 (0.6224) | -1.527 (0.589)
  LTA-RE, Wave III: Change at Week 22 (n= 2, 3, 2) | -0.116 (0.2867) | -0.549 (0.4627) | -1.239 (1.5038)
  LTA-RE, Wave V: Baseline (n= 2, 3, 3) | -0.567 (0.6834) | -0.792 (0.2929) | -1.19 (0.3631)
  LTA-RE, Wave V: Change at Week 22 (n= 2, 3, 3) | -0.474 (0.5435) | -0.214 (0.3107) | -1.237 (1.5458)
  LTA-LE, Wave I: Baseline (n= 2, 3, 4) | -0.918 (0.0708) | -0.875 (0.4212) | -1.445 (0.5468)
  LTA-LE, Wave I: Change at Week 22 (n= 2, 3, 3) | -0.409 (0.6445) | -0.268 (0.8163) | 0.078 (0.5695)
  LTA-LE, Wave III: Baseline (n= 2, 3, 4) | -1.602 (0.5149) | -1.057 (0.4761) | -1.643 (0.5086)
  LTA-LE, Wave III: Change at Week 22 (n= 2, 3, 3) | 0.265 (0.3271) | -0.374 (0.7773) | 0.053 (0.151)
  LTA-LE, Wave V: Baseline (n= 2, 3, 4) | -0.726 (0.5418) | -0.748 (0.2486) | -1.372 (0.5377)
  LTA-LE, Wave V: Change at Week 22 (n= 2, 3, 4) | -0.217 (0.4692) | -0.066 (0.2771) | 0.006 (0.3379)

24. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Square-root Transformed Latencies
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR square-root transformed latency (STL) by left and right ear were reported.
Time Frame: Baseline, Week 22
Population: ITT population.Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: square-root transformed (latency [ms])
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
square-root transformed (latency [ms])
  STL-RE, Wave I: Baseline (n= 3, 3, 3) | 1.312 (0.0886) | 2.03 (0.061) | 1.328 (0.0044)
  STL-RE, Wave I: Change at Week 22 (n= 3, 3, 3) | -0.002 (0.1734) | 0.08 (0.1935) | 0.145 (0.3167)
  STL-RE, Wave III: Baseline (n= 3, 3, 3) | 2.003 (0.1123) | 2.508 (0.0487) | 2.023 (0.0446)
  STL-RE, Wave III:Change at Week 22 (n= 3, 3, 2) | -0.021 (0.0884) | 0.056 (0.1593) | -0.008 (0.0107)
  STL-RE, Wave V: Baseline (n= 3, 3, 3) | 2.462 (0.0571) | 1.297 (0.091) | 2.461 (0.0461)
  STL-RE, Wave V: Change at Week 22 (n= 3, 3, 3) | -0.035 (0.0974) | 0.059 (0.1233) | 0.125 (0.2057)
  STL-LE, Wave I: Baseline (n= 3, 3, 4) | 1.315 (0.05) | 2.053 (0.055) | 1.332 (0.0858)
  STL-LE, Wave I: Change at Week 22 (n= 3, 3, 3) | -0.068 (0.0425) | -0.019 (0.1223) | 0.014 (0.0608)
  STL-LE, Wave III: Baseline (n= 3, 3, 4) | 2.012 (0.0805) | 2.522 (0.0464) | 2.04 (0.1236)
  STL-LE, Wave III: Change at Week 22 (n= 3, 3, 3) | -0.047 (0.0403) | -0.019 (0.0644) | 0.035 (0.0709)
  STL-LE, Wave V: Baseline (n= 3, 3, 4) | 2.473 (0.0559) | 1.26 (0.0824) | 2.5 (0.1208)
  STL-LE, Wave V: Change at Week 22 (n= 3, 3, 4) | -0.042 (0.0354) | 0.166 (0.0633) | 0.047 (0.0438)

25. Secondary Outcome: Change From Baseline in Auditory Brainstem Response (ABR) at Week 22: Square-root Transformed Amplitude
Description: ABR assessments were to be conducted under anesthesia and measured the electrical response evoked by acoustic stimuli as sound is processed along the auditory pathway. Data for change from baseline in ABR square-root transformed amplitude (STA) by left and right ear were reported.
Time Frame: Baseline, Week 22
Population: ITT population. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: square-root transformed(amplitude [mcV])
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Number analyzed (Participants) | 4 | 4 | 4
square-root transformed(amplitude [mcV])
  STA-RE, Wave I: Baseline (n= 2, 3, 3) | 0.7 (0.0303) | 0.644 (0.0896) | 0.507 (0.0933)
  STA-RE, Wave I: Week 22 (n= 2, 3, 3) | -0.193 (0.0535) | -0.172 (0.1615) | -0.044 (0.2298)
  STA-RE, Wave III: Baseline (n= 2, 3, 3) | 0.566 (0.1374) | 0.575 (0.171) | 0.479 (0.1274)
  STA-RE, Wave III: Week 22 (n= 2, 3, 2) | -0.038 (0.0838) | -0.122 (0.0927) | -0.211 (0.2317)
  STA-RE, Wave V: Baseline (n= 2, 3, 3) | 0.775 (0.2599) | 0.678 (0.1022) | 0.557 (0.0954)
  STA-RE, Wave V: Week 22 (n= 2, 3, 3) | -0.18 (0.2183) | -0.069 (0.1049) | -0.197 (0.2547)
  STA-LE, Wave I: Baseline (n= 2, 3, 4) | 0.632 (0.0224) | 0.655 (0.1437) | 0.499 (0.133)
  STA-LE, Wave I: Week 22 (n= 2, 3, 3) | -0.101 (0.1638) | -0.028 (0.1961) | 0.006 (0.1365)
  STA-LE, Wave III: Baseline (n= 2, 3, 4) | 0.456 (0.1162) | 0.601 (0.1508) | 0.45 (0.1131)
  STA-LE, Wave III: Week 22 (n= 2, 3, 3) | 0.057 (0.068) | -0.085 (0.1798) | 0.015 (0.0422)
  STA-LE, Wave V: Baseline (n= 2, 3, 4) | 0.709 (0.1896) | 0.692 (0.0873) | 0.518 (0.1488)
  STA-LE, Wave V: Week 22 (n= 2, 3, 4) | -0.084 (0.167) | -0.019 (0.0956) | -0.004 (0.0832)

ADVERSE EVENTS:
Time Frame: Baseline to Week 30 (follow-up)
Arm/Group | HGT-1410 10 mg | HGT-1410 45 mg | HGT-1410 90 mg
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGT-1410 10 mg (N=4) | HGT-1410 45 mg (N=4) | HGT-1410 90 mg (N=4)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device component issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medical device change (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HGT-1410 10 mg (N=4) | HGT-1410 45 mg (N=4) | HGT-1410 90 mg (N=4)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (5) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (6) | 1 (1) | 2 (2)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 1 (1)
Implant site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 2 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (5) | 2 (7) | 1 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (2)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 2 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CSF protein increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
CSF white blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Norovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (7)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Crying (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 0 (0) | 1 (11)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (7)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Labia enlarged (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infection prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Comparison to values obtained in a longitudinal, 12 month, natural history study of untreated participants with MPS IIIA was not reported as it was to be compared with another study protocol HGT-SAN-053 (NCT01047306).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.